CLINICAL TRIAL: NCT00979550
Title: The Effects of Aldara as an Adjunct to Laser Treatment of Port Wine Stains
Brief Title: The Effects of Aldara as an Adjunct to Laser Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to enroll enough participants
Sponsor: Henry Vasconez (Other)
Collaborators: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor-Investigator, Henry Vasconez, principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UK Aldara
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Port Wine Stains
Keywords: laser; pediatric; skin pigmentation
MeSH Terms: conditions — Hemangioma, Capillary; Pigmentation Disorders | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aldara cream (Experimental): Imiquimod (Aldara cream) will be applied nightly for four weeks after standard of care laser treatment for port wine stain.
  Interventions: Drug: Imiquimod
- non-medicated petroleum cream (Placebo Comparator): Non-medicated petroleum cream will be applied nightly for four weeks after standard of care laser treatment for port wine stain.
  Interventions: Drug: non-medicated petroleum cream

INTERVENTIONS:
Drug: Imiquimod — commercially available topical antiviral drug
  Other Names: Aldara
  Arms: Aldara cream
Drug: non-medicated petroleum cream — Over the counter topical cream used to aid the healing process in skin lesions
  Arms: non-medicated petroleum cream

SUMMARY:
The primary objective is to determine the effects of Aldara on the cosmetic outcome of laser treatment of vascular malformations.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blinded study. Volunteers who are scheduled for laser treatment of Port Wine Stains will be screened and eligible subjects will be asked to participate. The patients will be randomized and placed in the experimental or the control group. They will be given unlabeled sachets and instructed to apply the product each night to the right half of their treated lesion beginning the night after surgery for 4 weeks. Digital photographs of the Port Wine Stain will be taken prior to surgery and repeated at follow up appointments at 1 week, 1 month, 2 months, and 3 months after surgery. The photographs will be analyzed by blinded board certified plastic surgeons as well as a computer program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient between the ages of 2 and 60 years with a vascular malformation that is seeking cosmetic treatment.
* All races will be included as well as male and female.
* Clinical data on the usage of Aldara below the age of 2 years is limited and therefore all patients in the study will have to be at least 2 years of age.
* The majority of port wine stains are initially treated during childhood
* In order to determine the effectiveness of Aldara as an adjunct to laser therapy of Port Wine Stains, some of the patients in the study need to have lesions that have not undergone previous treatment.

Exclusion Criteria:

* Patients under the age of 2 or over the age of 60.
* Patients that have serious medical problems that would put them at risk of the anesthesia.
* Patients that have sensitivity reactions to the ingredients in the product including imiquimod, isostearic acid, cetyl alcohol, stearyl alcohol, white petrolatum, polysorbate 60, sorbitan monostearate, glycerin, xanthan gum, purified water, benzyl alcohol, methylparaben, and propylparaben.
* Patients who are pregnant or have significant immunodeficiency or autoimmune diseases.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Vasconez, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Division of Plastic Surgery, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aldara Cream: The patients will be randomized and placed in the experimental or the control group. They will be given unlabeled sachets and instructed to apply the product each night to the right half of their treated lesion beginning the night after surgery for 4 weeks. Digital photographs of the Port Wine Stain will be taken prior to surgery and repeated at follow up appointments at 1 week, 1 month, 2 months, and 3 months after surgery. The photographs will be analyzed by blinded board certified plastic surgeons as well as a computer program.
  Imiquimod (Aldara): .5 oz cream nightly to the affected area
- Non-medicated Petroleum Cream: The patients will be randomized and placed in the experimental or the control group. They will be given unlabeled sachets and instructed to apply the product each night to the right half of their treated lesion beginning the night after surgery for 4 weeks. Digital photographs of the Port Wine Stain will be taken prior to surgery and repeated at follow up appointments at 1 week, 1 month, 2 months, and 3 months after surgery. The photographs will be analyzed by blinded board certified plastic surgeons as well as a computer program.
  non-medicated petroleum cream: .5 oz cream nightly to the affected area
Period: Overall Study
Arm/Group | Aldara Cream | Non-medicated Petroleum Cream
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aldara Cream | Non-medicated Petroleum Cream | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Effects of Aldera Cream on the Reduction of Port Wine Stain (Vascular Malformation)
Description: Lesions will be digitally photographed and its surface area measured by blinded observers using image analysis software
Time Frame: 3 months
Arm/Group | Aldara Cream | Non-medicated Petroleum Cream
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Aldara Cream | Non-medicated Petroleum Cream
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No